CLINICAL TRIAL: NCT04925570
Title: Woebot for Substance Use Disorders Phase 2 RCT: Digitally Delivered Intervention for Reducing Problematic Substance Use
Brief Title: The Anchor Study: Digitally Delivered Intervention for Reducing Problematic Substance Use
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Woebot Health (Industry)
Collaborators: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 58725
Record Dates: First submitted 2021-05-25; First posted 2021-06-14 (Actual); Results first posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Alcohol Use Disorder (AUD); Substance Use Disorders
Keywords: Alcohol Use Disorder; Substance Use Disorder; AUD; SUD; AUD Treatment; SUD Treatment; Smartphone Application; Digital Therapeutic; Alcohol Use Disorder Treatment; Substance Use Disorder Treatment
MeSH Terms: conditions — Alcoholism; Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- W-SUDs (Experimental): Woebot (W-SUDs), a Conversational Agent (CA) instantaneously available 24 hours per day, 7 days per week, 'checks in' with users. Using conversational tones, it encourages mood tracking and delivers general psychoeducation as well as tailored empathy, cognitive behavior therapy (CBT)-based behavior change tools, and behavioral pattern insight. Woebot's app-based platform and user-centered design philosophy makes it an optimal modality for Substance Use Disorders (SUD) treatment delivery. It offers immediate, evidence-based tailored support in the patient's peak moment of craving.
  Interventions: Device: W-SUDs
- Digitally-delivered Psychoeducation (Other): Psychoeducation delivers weekly fact sheets that include information on:
  1. Alcohol-specific topics;
  2. Drug-specific topics;
  3. General addiction topics;
  4. Statistics relating to alcohol and substance use.
  Interventions: Other: Digitally-delivered Psychoeducation

INTERVENTIONS:
Device: W-SUDs — Woebot (W-SUDs) is an automated conversational agent, available through a smartphone application, that delivers evidence-based psychotherapeutics, empathy, and emotional health psychoeducation.
  Arms: W-SUDs
Other: Digitally-delivered Psychoeducation — A form of psychoeducation for those seeking treatment for their alcohol and/or substance use concern. Psychoeducation is commonly provided for those with substance use. Psychoeducation in substance use is intended to increase the users' knowledge of their substances of use, and effects on the body, behaviors, and consequences. The recipient of psychoeducation is expected to increase their own awareness of their substance use and ideally incorporate this newfound knowledge when making changes to their substance use. The information provided in this group are from factsheets found on NIAAA, NIDA, and CDC web pages.
  Arms: Digitally-delivered Psychoeducation

SUMMARY:
This study aims to validate W-SUDs as a digitally-delivered substance use disorder program through a fully-powered randomized control trial that will test the comparative efficacy of the mobile-app based substance use disorder program (W-SUDs) to reduce substance use relative to a psychoeducation control condition, which has no cognitive behavioral therapy and the content is not delivered through a conversational user interface.

DETAILED DESCRIPTION:
Phase II will evaluate the efficacy of W-SUDs in a large scale RCT relative to a psychoeducation control condition. Primary outcomes will be measures of the quantity and frequency of substance use including number of substance use occasions, heavy drinking days (if applicable) and percent reduction in substance use occasions. Additionally, Phase II will evaluate whether W-SUDs results in a greater reduction in substance-related problems compared to a psychoeducation control group and explore if engagement with W-SUDs, relative to psychoeducation control,

1. improves symptoms of depression and anxiety;
2. improves work productivity (i.e. reduce presenteeism/absenteeism);
3. reduces cravings;
4. improves situational confidence to resist substance use.

ELIGIBILITY:
Inclusion Criteria:

1. Have a smartphone
2. Endorse a substance use concern
3. Be between 18 and 65 years of age
4. Be available and committed to engage with the Woebot app
5. Be literate in English. (This is required for inclusion because all materials will be in English).

Exclusion Criteria:

1. Pregnancy (as W-SUDs will not be specifically developed to address the unique needs of this population)
2. Suicide attempt within the past year (12 months)
3. Symptoms of severe drug/alcohol history: History of delirium tremens; Experiencing hypertension, drenching sweats, seizures or confusion after stopping alcohol or drugs; Liver trouble (cirrhosis or hepatitis); Convulsions or GI bleeding due to drug/alcohol use
4. Opioid overdose within the past year (12 months)
5. Opioid misuse without medication-assisted treatment
6. Not residing in the U.S.
7. Previous Woebot use

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2022-11-14 (Actual); Primary Completion 2023-08-17 (Actual); Study Completion 2023-08-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith Prochaska, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

REFERENCES:
- [Derived] Moore JB, Chieng A, Pirner MC, Pajarito S, Vogel EA, Bowdring MA, Bullard L, Robinson A, Prochaska JJ. Mitigating fraud in a fully decentralized clinical trial of a digital health intervention. Ann Behav Med. 2025 Jan 4;59(1):kaaf047. doi: 10.1093/abm/kaaf047. PMID 40548528
- [Derived] Prochaska JJ, Vogel EA, Chieng A, Baiocchi M, Pajarito S, Pirner M, Darcy A, Robinson A. A relational agent for treating substance use in adults: Protocol for a randomized controlled trial with a psychoeducational comparator. Contemp Clin Trials. 2023 Apr;127:107125. doi: 10.1016/j.cct.2023.107125. Epub 2023 Feb 20. PMID 36813084

RESULTS

PARTICIPANT FLOW:
Groups:
- Digitally-delivered Psychoeducation: Psychoeducation delivers weekly fact sheets that include information on:
  1. Alcohol-specific topics;
  2. Drug-specific topics;
  3. General addiction topics;
  4. Statistics relating to alcohol and substance use.
  Digitally-delivered Psychoeducation: A form of psychoeducation for those seeking treatment for their alcohol and/or substance use concern. Psychoeducation is commonly provided for those with substance use. Psychoeducation in substance use is intended to increase the users' knowledge of their substances of use, and effects on the body, behaviors, and consequences. The recipient of psychoeducation is expected to increase their own awareness of their substance use and ideally incorporate this newfound knowledge when making changes to their substance use. The information provided in this group are from factsheets found on NIAAA, NIDA, and CDC web pages.
Period: Overall Study
Arm/Group | W-SUDs | Digitally-delivered Psychoeducation
Started | 131 | 127
Completed | 107 | 95
Not Completed | 24 | 32
Not completed — Protocol Violation | 24 | 30
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | W-SUDs | Digitally-delivered Psychoeducation | Total
Number analyzed (Participants) | 107 | 95 | 202
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.2 (11.4) | 38.6 (9.2) | 38.3 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 58 | 108
  Male | 57 | 37 | 94
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 11 | 23
  Not Hispanic or Latino | 94 | 84 | 178
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 17 | 28 | 45
  White | 86 | 58 | 144
  More than one race | 0 | 3 | 3
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 107 | 95 | 202
Gender [Count of Participants; unit: Participants]
  Woman | 50 | 56 | 106
  Man | 56 | 37 | 93
  Non-binary | 1 | 2 | 3
Sexual Orientation [Count of Participants; unit: Participants]
  Heterosexual | 90 | 84 | 174
  Gay or Lesbian | 8 | 2 | 10
  Bisexual | 5 | 5 | 10
  Queer | 0 | 1 | 1
  Pansexual | 2 | 3 | 5
  Don't know | 2 | 0 | 2
Marital Status [Count of Participants; unit: Participants]
  Married/Cohabitating/Partnered | 53 | 52 | 105
  Divorced/Separated/Widowed | 13 | 9 | 22
  Never married/Single | 41 | 34 | 75
Educational Degree [Count of Participants; unit: Participants]
  High School Degree or Less | 17 | 13 | 30
  Some College/Technical School | 37 | 36 | 73
  College Degree | 30 | 27 | 57
  Graduate or Post-graduate Degree | 23 | 19 | 42
Employment Status [Count of Participants; unit: Participants]
  Employed Part or Full-Time | 74 | 61 | 135
  Unemployed (homemaker, student, retired) | 33 | 34 | 67
Disability Status [Count of Participants; unit: Participants]
  Yes (has a disability) | 8 | 10 | 18
  No (does not have a disability) | 98 | 85 | 183
  Prefer not to answer | 1 | 0 | 1
Insurance Status [Count of Participants; unit: Participants]
  Private | 56 | 47 | 103
  Medicaid or Medicare | 32 | 33 | 65
  TRICARE | 0 | 2 | 2
  VA | 1 | 1 | 2
  Doesn't have insurance | 18 | 10 | 28
  Prefer not to answer | 0 | 2 | 2
Lifetime Mental Health Condition [Number; unit: participants]
  Unipolar Depression | 20 | 26 | 48
  Bipolar/Manic Depression | 9 | 5 | 14
  Anxiety Disorder | 34 | 32 | 66
  Substance Use Disorder | 8 | 7 | 15
  Other Mental Health Disorder | 23 | 24 | 47
  Multiple Diagnoses | 29 | 26 | 55
  No History of Mental Illness | 62 | 48 | 111
Prior Therapy Experience [Count of Participants; unit: Participants]
  Never in Therapy | 66 | 52 | 118
  Formerly in Therapy | 28 | 25 | 53
  Currently in Therapy | 13 | 18 | 31
Psychiatric Medications [Count of Participants; unit: Participants]
  Currently Taking Psychiatric Medications | 25 | 17 | 42
  Not Currently Taking Psychiatric Medications | 82 | 78 | 160
Past 30 Day SUD Treatment [Count of Participants; unit: Participants]
  Self-help Groups | 2 | 5 | 7
  Outpatient Services | 5 | 5 | 10
  Intensive Outpatient/Residential | 2 | 2 | 4
  No Treatment | 98 | 83 | 181
Past 30 Day Medication Use for SUD Treatment [Count of Participants; unit: Participants]
  Yes (Used medication) | 2 | 1 | 3
  No (Did not use medication) | 105 | 94 | 199
Primary, Secondary, or Tertiary Problematic Substance [Number; unit: participants]
  Alcohol | 76 | 72 | 148
  Cannabis | 27 | 35 | 62
  Stimulants | 20 | 15 | 35
  Cocaine | 16 | 9 | 25
  Tobacco | 36 | 34 | 70
  Other (e.g., Heroin, Hallucinogens, Inhalants) | 22 | 15 | 37

OUTCOME MEASURES:

1. Primary Outcome: Change in Number of Substance Use Occasions
Description: Change in number of substance use occasions in the past 30 days
Time Frame: Change from Baseline to Mid-treatment at 4 weeks; Change from Baseline to Post-treatment at 8 weeks; Change from Baseline to Follow-up at 12 weeks
Measure: Mean (Standard Deviation); unit: occasions
Arm/Group | W-SUDs | Digitally-delivered Psychoeducation
Number analyzed (Participants) | 107 | 95
occasions
  Week 4 | -11.3 (15.9) | -11.2 (12.9)
  Week 8 | -13.6 (15.4) | -12.9 (15.3)
  Week 12 | -15.7 (18) | -15.4 (16.6)

2. Secondary Outcome: Drug Abuse Screening Test (DAST-10)
Description: Measure of drug abuse related consequences. The DAST-10 is a brief, 10-item self-report measure that assesses consequences related to drug abuse, excluding alcohol and tobacco. The range is 0-10, where higher scores indicate greater severity. Adapted from past 12 months to past 30 days.
Time Frame: Change from Baseline to Post-treatment at 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | W-SUDs | Digitally-delivered Psychoeducation
Number analyzed (Participants) | 65 | 54
score on a scale | -1.21 (2.33) | -1.95 (1.99)

3. Secondary Outcome: Working Alliance Inventory (WAI-SR)
Description: Measure of working alliance. A measure of therapeutic alliance that assesses three key aspects of the therapeutic alliance: (a) agreement on the tasks of therapy, (b) agreement on the goals of therapy and (c) development of an affective bond. Task, goal, and bond subscales scores range from 5-20, with higher scores indicating greater alliance. The present study utilized the validated 12-item Short-Revised version (WAI-SR) with minor changes to language, replacing "therapist" with "Woebot".
Time Frame: Post-treatment at 8 weeks
Population: Number analyzed for each subscale differs from the overall number analyzed due to missingness.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | W-SUDs
Number analyzed (Participants) | 98
score on a scale
  Goal: number analyzed (Participants) | 97
  Goal | 14.8 (4.4)
  Task | 14.4 (4.5)
  Bond: number analyzed (Participants) | 97
  Bond | 15.2 (4.5)

4. Secondary Outcome: Stanford Presenteeism Scale (SPS-6)
Description: Measure of the effects of substance use on productivity. The SPS-6 is a 6-item self-report measure used to assess perceptions of the effects of substance use on past 2-week work productivity. Response options range from strongly disagree (1) to strongly agree (5). Total scores range from 6 to 30, where higher scores indicate higher presenteeism.
Time Frame: Change from Baseline to Post-treatment at 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | W-SUDs | Digitally-delivered Psychoeducation
Number analyzed (Participants) | 72 | 61
score on a scale | -5.42 (7.2) | -4.12 (6.97)

5. Secondary Outcome: Thoughts About Abstinence (TAA): Desire to Quit, Expected Success at Quitting, Expected Difficulty of Quitting Items
Description: Modified for alcohol and substances. 4-item questionnaire assessing desire to quit, expected success at quitting, expected difficulty of quitting, and goal. Each of the first three items is rated on a scale of 1 to 10 where 1 is the lowest (desire, expectation, confidence) and 10 is the highest (desire, expectation, confidence). The scores are not combined. Goal for use is a single response selection item, with the option to provide a text explanation if none of the goals align. Goal data are reported as a separate outcome measure.
Time Frame: Change from Baseline to Post-treatment at 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | W-SUDs | Digitally-delivered Psychoeducation
Number analyzed (Participants) | 107 | 95
score on a scale
  Desire to quit | 0.21 (2.33) | 0.12 (2.71)
  Expected success at quitting | 0.42 (2.37) | 0.53 (2.72)
  Expected difficulty of quitting | -0.64 (2.44) | -0.28 (2.91)

6. Secondary Outcome: Thoughts About Abstinence (TAA): Goal Item
Description: Modified for alcohol and substances. 4-item questionnaire assessing desire to quit, expected success at quitting, expected difficulty of quitting, confidence in ability to quit, and goal. Each of the first three items is rated on a scale of 1 to 10 where 1 is the lowest (desire, expectation, confidence) and 10 is the highest (desire, expectation, confidence). The scores are not combined. Goal for use is a single response selection item, with the option to provide a text explanation if none of the goals align. Desire to Quit, Expected Success at Quitting, Expected Difficulty of Quitting item data are reported as a separate outcome measure.
Time Frame: Baseline and Post-treatment at 8 weeks
Population: Number analyzed in categories reported at 8 weeks differs from overall number analyzed due to data missingness.
Measure: Number; unit: participants
Arm/Group | W-SUDs | Digitally-delivered Psychoeducation
Number analyzed (Participants) | 107 | 95
participants
  No goal (Baseline) | 10 | 12
  Controlled use (Baseline) | 25 | 22
  Short-term abstinence (Baseline) | 14 | 9
  Occasional use when there is urge (Baseline) | 17 | 19
  Quit, but might slip (Baseline) | 13 | 11
  Quit forever (Baseline) | 25 | 18
  Other (Baseline) | 3 | 4
  No goal (8 weeks): number analyzed (Participants) | 100 | 90
  No goal (8 weeks) | 16 | 12
  Controlled use (8 weeks): number analyzed (Participants) | 100 | 90
  Controlled use (8 weeks) | 19 | 28
  Short-term abstinence, then decide about continued use (8 weeks): number analyzed (Participants) | 100 | 90
  Short-term abstinence, then decide about continued use (8 weeks) | 15 | 6
  Occasional use when there is urge (8 weeks): number analyzed (Participants) | 100 | 90
  Occasional use when there is urge (8 weeks) | 8 | 6
  Quit, but might slip (8 weeks): number analyzed (Participants) | 100 | 90
  Quit, but might slip (8 weeks) | 14 | 11
  Quit forever (8 weeks): number analyzed (Participants) | 100 | 90
  Quit forever (8 weeks) | 25 | 21
  Other (8 weeks): number analyzed (Participants) | 100 | 90
  Other (8 weeks) | 3 | 5
  Prefer not to answer (8 weeks): number analyzed (Participants) | 100 | 90
  Prefer not to answer (8 weeks) | 0 | 1

7. Secondary Outcome: Usage Rating Profile - Intervention (URPI)-Acceptability
Description: Measure of acceptability. A 9-item subscale that inquires about intervention acceptability. For the purposes of this study, an adapted 6-item version of the subscale was utilized. Items are rated on a 6-point Likert scale (1 = "strongly disagree" to 6 = "strongly agree"). Total acceptability scores range from 6-36, with higher scores indicating greater intervention acceptability.
Time Frame: Post-treatment at 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | W-SUDs | Digitally-delivered Psychoeducation
Number analyzed (Participants) | 99 | 89
score on a scale | 30.1 (5.6) | 30.3 (5.8)

8. Secondary Outcome: Usage Rating Profile - Intervention (URPI)-Feasibility
Description: Measure of feasibility. A 6-item subscale that inquires about factors that impact treatment usage (i.e., intervention quality). Items are rated on a 6-point Likert scale (1 = "slightly disagree" to 6 = "strongly agree"). Total feasibility scores range from 6-36, with higher scores indicating greater intervention feasibility.
Time Frame: Post-treatment at 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | W-SUDs | Digitally-delivered Psychoeducation
Number analyzed (Participants) | 99 | 89
score on a scale | 28.0 (3.5) | 29.8 (2.6)

9. Secondary Outcome: Client Satisfaction Questionnaire (CSQ-8)
Description: Measure of satisfaction. An 8-item measure used to assess client's satisfaction with treatment on a 4-point scale. Example questions include, "How would you rate the quality of service you received"? and "Did you get the kind of service you wanted?" Total sums range from 8-32, with high scores indicating greater satisfaction with the W-SUDs mobile application.
Time Frame: Post-treatment at 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | W-SUDs | Digitally-delivered Psychoeducation
Number analyzed (Participants) | 99 | 87
score on a scale | 26.9 (5.2) | 28.1 (4.5)

10. Secondary Outcome: Short Inventory of Problems- Alcohol and Drugs (SIP-AD)
Description: The SIP-AD assesses substance use problems in the past 30 days. The scored variables, total scores and 15-item mean, summarize consequences of alcohol and drug use. Scores range from 0-45, where greater scores indicate greater substance use problems.
Time Frame: as for outcome 1
Population: Number analyzed for each timepoint differs from the overall number analyzed due to missingness.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | W-SUDs | Digitally-delivered Psychoeducation
Number analyzed (Participants) | 100 | 93
score on a scale
  Mid-treatment at 4 weeks: number analyzed (Participants) | 98 | 91
  Mid-treatment at 4 weeks | -8.02 (9.35) | -7.39 (9.95)
  Post-treatment at 8 weeks: number analyzed (Participants) | 100 | 90
  Post-treatment at 8 weeks | -9.02 (11.6) | -9.24 (10.2)
  Follow-up at 12 weeks: number analyzed (Participants) | 98 | 93
  Follow-up at 12 weeks | -11.5 (11.5) | -10.9 (11.5)

11. Secondary Outcome: Patient Health Questionnaire (PHQ-8)
Description: Measure of depression severity. An 8-item abbreviated version of the PHQ-9 used to assess mood symptoms. The PHQ-8 excludes an item assessing suicidality. Items are rated on a 4-point Likert scale (0 = "not at all" to 3 = "nearly every day"). Total score between 0-24, with higher scores indicating greater severity of depression symptoms.
Time Frame: as for outcome 1
Population: Number analyzed for each timepoint differs from the overall number analyzed due to missingness.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | W-SUDs | Digitally-delivered Psychoeducation
Number analyzed (Participants) | 100 | 93
score on a scale
  Mid-treatment at 4 weeks: number analyzed (Participants) | 98 | 91
  Mid-treatment at 4 weeks | -1.84 (4.24) | -1.44 (4.45)
  Post-treatment at 8 weeks: number analyzed (Participants) | 100 | 90
  Post-treatment at 8 weeks | -2.82 (4.65) | -2.05 (5.95)
  Follow-up at 12 weeks: number analyzed (Participants) | 98 | 93
  Follow-up at 12 weeks | -2.83 (4.79) | -2.87 (6.3)

12. Secondary Outcome: Generalized Anxiety Disorder (GAD-7)
Description: Measure of anxiety severity. A 7-item self-report measure used to assess the frequency and severity of anxious thoughts and behaviors over the past 2 weeks. Items are rated on a 4-point Likert scale (0 = "not at all" to 3 = "nearly every day").Total scores range from 0-21, where higher scores indicate greater severity of anxiety symptoms.
Time Frame: as for outcome 1
Population: Number analyzed for each timepoint differs from the overall number analyzed due to missingness.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | W-SUDs | Digitally-delivered Psychoeducation
Number analyzed (Participants) | 100 | 93
score on a scale
  Mid-treatment at 4 weeks: number analyzed (Participants) | 98 | 91
  Mid-treatment at 4 weeks | -1.31 (4.05) | -1.56 (3.97)
  Post-treatment at 8 weeks: number analyzed (Participants) | 100 | 90
  Post-treatment at 8 weeks | -1.88 (4.77) | -1.72 (4.91)
  Follow-up at 12 weeks: number analyzed (Participants) | 98 | 93
  Follow-up at 12 weeks | -2.09 (4.67) | -2.57 (5.08)

13. Secondary Outcome: Brief Situational Confidence Questionnaire (BSCQ)
Description: Measure of self-confidence. The 8-item BSCQ is a state dependent measure that assesses self-confidence to resist the urge to drink heavily or use drugs in a variety of situations. Each of the 8 scale situations consists of a 100-mm line, anchored by 0% ("not at all confident") and 100% ("totally confident") where clients are asked to indicate confidence on a scale from 0% to 100%. Higher scores are associated with greater confidence.
Time Frame: as for outcome 1
Population: Number analyzed for each timepoint differs from the overall number analyzed due to missingness.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | W-SUDs | Digitally-delivered Psychoeducation
Number analyzed (Participants) | 96 | 90
score on a scale
  Mid-treatment at 4 weeks: number analyzed (Participants) | 95 | 88
  Mid-treatment at 4 weeks | 7.3 (21.4) | 10.4 (23.2)
  Post-treatment at 8 weeks: number analyzed (Participants) | 96 | 86
  Post-treatment at 8 weeks | 6.77 (20.4) | 11.6 (20.3)
  Follow-up at 12 weeks: number analyzed (Participants) | 94 | 90
  Follow-up at 12 weeks | 11.6 (21.8) | 15.6 (26.1)

14. Secondary Outcome: Craving Ratings
Description: Self-reported ratings of craving intensity. Craving is assessed with a single question, "In the past 7 days, how much were you bothered by cravings or urges to drink alcohol or use drugs?". The question is rated on a scale of 0 to 4 where 0 = not at all, 1 = a little bit, 2 = moderately, 3 = quite a bit, and 4 = extremely. Greater scores indicate a more intense urge to use.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | W-SUDs | Digitally-delivered Psychoeducation
Number analyzed (Participants) | 107 | 95
score on a scale
  Mid-treatment at 4 weeks | -0.418 (0.994) | -0.56 (1.14)
  Post-treatment at 8 weeks | -0.66 (1.18) | -0.722 (1.2)
  Follow-up at 12 weeks | -0.816 (1.15) | -0.892 (1.4)

15. Secondary Outcome: Past Month Number of Binge Days
Description: Assessed with the Quick Drinking Screen (QDS), a measure of alcohol consumption. The QDS is a brief self-report measure used to assess average alcohol consumption over a specified time period (in the present study it was the past 30 days). The QDS collects drinking data for three variables including number of days drinking, number of standard drinks per drinking day, and number of binge/risky drinking days. Binge/risky drinking days is defined as days when they have had 5 or more standard drinks (for men) or 4 or more standard drinks (for women).
Time Frame: as for outcome 1
Population: Number analyzed for each timepoint differs from the overall number analyzed due to missingness.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | W-SUDs | Digitally-delivered Psychoeducation
Number analyzed (Participants) | 78 | 67
days
  Mid-treatment at 4 weeks: number analyzed (Participants) | 78 | 64
  Mid-treatment at 4 weeks | -4.26 (6.88) | -2.45 (5.66)
  Post-treatment at 8 weeks: number analyzed (Participants) | 75 | 67
  Post-treatment at 8 weeks | -4.09 (6.35) | -2.51 (6.02)
  Follow-up at 12 weeks: number analyzed (Participants) | 70 | 63
  Follow-up at 12 weeks | -5.43 (7.21) | -3.14 (7.75)

16. Secondary Outcome: Past Month Average Standard Drinks in a Week
Description: Assessed with the Quick Drinking Screen (QDS), a measure of alcohol consumption. The QDS is a brief self-report measure used to assess average alcohol consumption over a specified time period (in the present study it was the past 30 days). The QDS collects drinking data for three variables including number of days drinking, number of standard drinks per drinking day, and number of binge/risky drinking days. Binge/risky drinking days is defined as days when they have had 5 or more standard drinks (for men) or 4 or more standard drinks (for women). Number of standard drinks per week is calculated by multiplying number of standard drinks per day in the past month and number of binge days per month.
Time Frame: as for outcome 1
Population: Number analyzed for each timepoint differs from the overall number analyzed due to missingness.
Measure: Mean (Standard Deviation); unit: Drinks per week
Arm/Group | W-SUDs | Digitally-delivered Psychoeducation
Number analyzed (Participants) | 78 | 67
Drinks per week
  Mid-treatment at 4 weeks: number analyzed (Participants) | 78 | 64
  Mid-treatment at 4 weeks | -7.62 (14.9) | -6.92 (12.4)
  Post-treatment at 8 weeks: number analyzed (Participants) | 75 | 67
  Post-treatment at 8 weeks | -8.67 (14.7) | -8.18 (11.5)
  Follow-up at 12 weeks: number analyzed (Participants) | 70 | 63
  Follow-up at 12 weeks | -11.1 (15.7) | -9.43 (13.9)

ADVERSE EVENTS:
Time Frame: Serious adverse events were assessed at post-treatment and follow-up at 8-weeks and 12-weeks from baseline, respectively.
Description: Serious adverse events occurring during treatment were assessed for hospitalization related to substance use, suicide attempt, alcohol or drug overdose, and severe withdrawal (e.g., delirium tremens). Positive endorsements were followed up with questions about the timing, diagnosis, and resolution. If additional details were needed to determine whether the event was study related, a team member reached out to the participant.
Arm/Group | W-SUDs | Digitally-delivered Psychoeducation
All-Cause Mortality (participants affected / at risk) | 0/107 | 0/95
Serious Adverse Events (participants affected / at risk) | 0/107 | 0/95
Other Adverse Events (participants affected / at risk) | 0/107 | 0/95

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2023-03-17): https://cdn.clinicaltrials.gov/large-docs/70/NCT04925570/Prot_008.pdf
  • Statistical Analysis Plan (2023-03-17): https://cdn.clinicaltrials.gov/large-docs/70/NCT04925570/SAP_009.pdf
  • Informed Consent Form (2023-03-17): https://cdn.clinicaltrials.gov/large-docs/70/NCT04925570/ICF_007.pdf